CLINICAL TRIAL: NCT03095703
Title: Sirolimus for the Treatment of Severe Intestinal Polyposis in Patients With Familial Adenomatous Polyposis (FAP): a Pilot Study
Brief Title: Sirolimus and Familial Adenomatous Polyposis (FAP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Professor MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL55868.018.15
Record Dates: First submitted 2017-03-21; First posted 2017-03-30 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-08

CONDITIONS: Adenomatous Polyposis Coli
Keywords: Sirolimus; Intestinal adenomas
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: A Prospective phase II pilot study with 5 patients with a follow-up of 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sirolimus (Experimental): All patients will receive sirolimus for the duration of the study, with a trough level target range of 5-8 ng/ml.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Participants will be given sirolimus tablets. The starting dose is 2 mg once daily which will be given in 1mg tablets. On day 7 the first trough level is measured (using the LC-MS/MS method) and if not within the target range of 5-8ng/ml, dosing adjustments are made. In case of dosing adjustments, the next trough level is measured seven days later and this is repeated weekly until the target range is achieved. In case trough levels are within the target range, the next trough level measurement is at month 3, after which dosing adjustments are made if necessary, and at month 6. The maximum daily dose is 40mg. No placebo is given.
  Other Names: Rapamune

SUMMARY:
The aim of the study is to investigate the effect of sirolimus on the progression of intestinal adenomas in patients with FAP and to assess the safety of this treatment.

DETAILED DESCRIPTION:
SUMMARY Rationale: Due to the presence of numerous colorectal polyps, nearly all patients with familial adenomatous polyposis (FAP) develop colorectal cancer (CRC) at an average age of 45 years, if left untreated. Therefore, a prophylactic colectomy is recommended. After surgery, adenomas are likely to reappear in the pouch or rectum. Recently, studies in APC-deficient mice have shown that the mTOR inhibitor sirolimus can cause intestinal tumour cells to undergo growth arrest and differentiation and could even lead to regression of polyps. In current practice, sirolimus is used as an immunomodulator for patients after renal transplantation. Sirolimus has never been investigated in patients with FAP. The hypothesis of the study is that sirolimus could lead to regression of intestinal polyps in patients with FAP.

Objective: The aim of the study is to investigate the effect of sirolimus on the progression of intestinal adenomas in patients with FAP and to assess the safety of this treatment.

Study design: A prospective phase II pilot study with a follow-up of 6 months. Study population: Five patients with FAP will be selected and invited for study participation. Patients need to be 18 years or older, have a genetically confirmed APC mutation with a classical FAP phenotype and a subtotal colectomy with an ileo-rectal anastomosis (IRA) or a total colectomy with an ileo-anal pouch anastomosis (IPAA) with severe polyposis.

Intervention: All patients will receive sirolimus for the duration of the study, with a trough level target range of 5-8 ng/ml.

Main study parameters/endpoints: The main study parameters are the effect of sirolimus on the size of 5 marked polyps and safety of this treatment. Safety outcomes will be assessed by summary analysis of adverse events, clinical laboratory abnormalities and regular physical examination. Additional parameters are the effect on the number of polyps, global polyp burden, histopathology and patient-reported quality of life. Cell proliferation and immunohistochemistry of mTOR targets in healthy intestinal mucosa and adenomatous tissue will be assessed.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: At baseline and at three monthly visits a medical history will be taken and physical examinations will be performed, as well as laboratory tests and HRQoL questionnaires. Trough level testing of sirolimus will be measured at day 7 after start of the study drug and weekly until the therapeutic range has been achieved, after which the next trough level will be measured at 3 and 6 months follow-up. Finally, monthly telephone check-ups will be carried out. LGI endoscopies will be done at baseline and at 6 months. For this study, patients are included with severe rectal or pouch polyposis as they are expected to have an indication for invasive surgery on a short-term base and no other less invasive alternative therapy is available.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* A genetically confirmed APC mutation
* Classical FAP phenotype (100-1000 colorectal adenomatous polyps)
* Subtotal colectomy with ileorectal anastomosis (IRA) or total colectomy with ileo-anal pouch anastomosis (IPAA)
* Severe rectal or pouch polyposis, defined as having >25 polyps amenable to complete removal (InSiGHT 2011 Staging System score of 3)
* Fertile patients must use effective contraception during study treatment and until 12 weeks after study treatment

Exclusion Criteria:

* Inability to give informed consent
* Participation in another interventional clinical trial
* Subjects who are pregnant or breast-feeding, proved with a negative pregnancy test if female of child-bearing potential
* Prior pelvic irradiation
* Invasive malignancy in the past 5 years
* Subjects who are HIV positive
* Subjects with severe systemic infections, current or within 2 weeks prior to study start
* Subjects with known severe restrictive or obstructive pulmonary disorders
* Known sucrase insufficiency, isomaltase insufficiency, fructose intolerance, glucose malabsorption, galactose malabsorption, galactose intolerance or Lapp-lactase deficiency
* History of pulmonary embolism or deep venous thrombosis
* Major surgery less than or equal to 2 weeks prior to enrollment or any planned surgery within treatment period
* Active post-operative complication, e.g. infection, delayed wound healing
* History of hypersensitivity to sirolimus or to drugs of similar chemical classes
* Regular NSAID use (defined as more than twice a week for 4 consecutive weeks) within 3 months prior to baseline
* Use of other FAP directed drug therapies (accepted if discontinued 3 months prior to start of the study)
* Subjects requiring systemic anticoagulation
* Co-medication that could interact with sirolimus
* Abnormal laboratory results (assessed within 14 days prior to start of study drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Dekker, MD, PhD, Principal Investigator — Academic Medical Centre Amsterdam
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roos VH, Meijer BJ, Kallenberg FGJ, Bastiaansen BAJ, Koens L, Bemelman FJ, Bossuyt PMM, Heijmans J, van den Brink G, Dekker E. Sirolimus for the treatment of polyposis of the rectal remnant and ileal pouch in four patients with familial adenomatous polyposis: a pilot study. BMJ Open Gastroenterol. 2020 Dec;7(1):e000497. doi: 10.1136/bmjgast-2020-000497. PMID 33376109

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patients with Familial Adenomatous Polyposis syndrome.
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [42 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Marked Polyp Size
Description: Effect of sirolimus on the size of 5 marked polyps per patient based on video observations.
Time Frame: 6 Months
Measure: Number; unit: Size of marked polyps
Units Other Than Participants: Size of marked polyps
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Number analyzed (Size of marked polyps) | 20
Size of marked polyps
  Decrease in marked polyp size | 16
  Same marked polyp size | 4
  Increase in marked polyp size | 0

2. Primary Outcome: Median Number of Treatment-Related Adverse Events Per Participant
Description: Summary analysis of adverse events, clinical laboratory abnormalities and regular physical examination.
Time Frame: 6 Months
Measure: Median (Full Range); unit: Number of Adverse Events
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Number of Adverse Events | 10 [4 to 16]

3. Secondary Outcome: Median Difference in Number of Intestinal Polyps
Description: Number of intestinal polyps was determined by two independent reviewers, blinded for the order of videos (before and after treatment). The median difference comparing baseline en after 6 months of treatment was reported.
Time Frame: 6 Months
Measure: Median (Full Range); unit: Median number of polyps
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Median number of polyps | 25.75 [6.5 to 50]

4. Secondary Outcome: Global Polyp Burden
Description: The global polyp burden is estimated by the endoscopist and two independent reviewers. The second video in the pair could take the value of -2 (much better), -1 (better), 0 (same), 1 (worse) or 2 (much worse) relative to the first video. Mean scores are calculated for each subject and averaged for the three reviewers. If the assessment of the reviewers differs by more than 1 point from the assessment of the endoscopist, consensus is needed.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Participants
  Much better | 0
  Better | 3
  Same | 1
  Worse | 0
  Much worse | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The primary objective was to assess the safety outcomes by analysis of adverse events (by monthly telephone calls), laboratory abnormalities and regular physical examination (during hospital visits at 3 and 6 months).
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=4)
Desmoid tumor (Musculoskeletal and connective tissue disorders) | 1 (1) — Discovery of a desmoid tumour in the abdominal wall (2.7 × 1.7 × 8.0cm) located near a scar.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=4)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (14) — 29% had gastrointestinal disorders.
Skin problems (Skin and subcutaneous tissue disorders) | 3 (5) — 12% had skin disorders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03095703/Prot_SAP_000.pdf